CLINICAL TRIAL: NCT01371760
Title: Randomized Multi-centered Study for Evaluating the Efficacy and Safety of Angioplastic Surgery of the Extracranial Veins in the Treatment of Multiple Sclerosis. Studio Randomizzato Multicentrico Per la Valutazione Dell'Efficacia e Sicurezza Dell'Intervento di Disostruzione Delle Vene Extracraniche Nel Trattamento Della Sclerosi Multipla
Brief Title: BRAVE-DREAMS (BRAin VEnous DRainage Exploited Against Multiple Sclerosis)
Acronym: BRAVE-DREAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S. Anna Hospital (Other)
Collaborators: Regione Emilia-Romagna (Other)
Responsible Party: Principal Investigator, Paolo Zamboni, PI, S. Anna Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S. Anna Hospital
Record Dates: First submitted 2011-06-07; First posted 2011-06-13 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Sclerosis; Venous Insufficiency
Keywords: Multiple sclerosis; Chronic cerebrospinal venous insufficiency; Percutaneous Transluminal Angioplasty (PTA); Internal jugular vein; Azygous vein
MeSH Terms: conditions — Multiple Sclerosis; Venous Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The patients will undergo PTA of the extracranial cerebral veins
  Interventions: Procedure: Venous PTA
- Controls (Sham Comparator): The patients will undergo sham procedure
  Interventions: Other: Catheter Venography

INTERVENTIONS:
Procedure: Venous PTA — PTA of the internal jugular and/or azygous vein
  Arms: Intervention
Other: Catheter Venography — The patients will undergo catheter venography but not PTA
  Arms: Controls

SUMMARY:
To assess in a double blinded randomized control trial (RCT) study design safety and effectiveness of balloon angioplasty of the main extracranial and extravertebral veins in multiple sclerosis (MS) associated to chronic cerebrospinal venous insufficiency (CCSVI).

Mean follow-up 1 year. 5-8 Italian centres 360 relapsing remitting (RR) MS patients will be randomized, with expanded disability disease scale (EDSS) ranging 2-5.5, age 18-65.

DETAILED DESCRIPTION:
Safety will be assessed by measuring serious and minor adverse effects related to treatment.

Effectiveness will be assessed by measuring 2 primary endpoints:

1. Clinical parameters will be expressed in an integrated functional measure leading to the score, respectively, of improved, stable, worsened. Functional assessment is performed by tools permitting a quantification and will be made by a team of independent assessors. Clinical instrumental evaluation will be performed at baseline, and subsequently on 3 months basis. The outcome parameters leading to the composite functional measure are instrumental parameters, less assessor dependent, singularly validated for measuring the disability in MS. They are the followings: A) Dynamic Balance Assessment: Balance Master Limits of Stability (LOS). In static platform, swinging to reach the set position of center of pressure. B) Walking Function: The subject walks spontaneously for 10 meters with chronometric measure of time counting the number of steps. The test calculates the walk ratio i.e. ratio between length and step frequency. C) Manual dexterity. Box & Block test, moving wooden cubes. D) Sphincter control: Post-voiding residual by ultrasounds. F) Visual acuity: Low-contrast visual acuity Sloan Letter Chart.
2. Magnetic Resonance Imaging (MRI) outcome measures: T1Gad active lesion.T2 lesion volume MRI evaluation at baseline, 6, 12 months.

Secondary endpoints are: EDSS, chronic fatigue, cognitive function, rate of restenosis, annualized relapse rate.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by CCSVI associated with MS
* relapsing-remitting and\or secondary progressive
* 18-65 years old
* EDSS 2-5
* disease duration < 10y
* No relapse in the 30 days preceding the procedure
* clinical stability in the last 6 months with disease mod. treatments
* Patients under the best available therapy

Exclusion Criteria:

* patients previously treated for CCSVI or inserted in other clinical trials in the last 3 months
* under treatment with natalizumab
* pregnant or refusing to adopt contraception
* presence of significant comorbidities
* alcool-drug abuse
* thrombophilia
* contraindication to MR

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical parameters in an integrated functional score | Baseline; 12 months
  Five neurological parameters will be measured by the means of proper validated tools along 1 year of follow-up. The evaluation leads to a score, respectively expressed as improved, stable, fluctuant, worsened.
MRI outcome measures: T1Gad active lesion.T2 lesion volume MRI evaluation. | Baseline; 12 months
  Standard MRI parameters will be assessed by the means of a blinded centre of lecture. Outcome measurement will be performed at baseline, 6 months and at 1 year follow-up.

SECONDARY OUTCOMES:
EDSS | Baseline; 12 months
  EDSS will be assessed along 1 year follow-up.
Chronic fatigue | Baseline; 12 months
  This highly disabling symptom completely orphan of effective therapy will be measured by M-FIS (Modified-Fatigue Impact Scale).
Cognitive function | Baseline; 12 months
  Cognitive functions will be measured by the means of MoCA mental state questionnaire.
Annualized relapse rate | Baseline; 12 months
  In the sub population affected by the RR clinical form the number of relapse will be assessed.
Patency rate | Baseline; 12 months
  The rate of successful PTA will be assessed by the means of postoperative Doppler sonography.
Emotional status | Baseline; 1 year
  Anxiety and Depression Scale for use with multiple sclerosis patients will be administered.
Memory and cognition | Baseline; 1 year
  The assessment will be performed by the means of PASAT - Paced Auditory Serial Addition Test
Overactive Bladder | Baseline; 1 year
  Overactive Bladder symptom will be measured by the means of validated Overactive Bladder Questionnaire-b.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Zamboni, MD, Principal Investigator — S. Anna Hospital, University of Ferrara, Ferrara, Italy; Graziella Filippini, MD, Study Chair — Istituto Neurologico Besta, Milano, Italy
Locations (2):
- Italy (2):
  - S. Anna Hospital, Ferrara, Fe
  - S. Anna Hospital, University of Ferrara, Ferrara, Italy, Ferrara

IPD SHARING:
Plan to Share IPD: Yes
Data analysis on behalf of the independent Biostatistic Center will be completed within May 2016

REFERENCES:
- [Result] Zamboni P, Galeotti R, Menegatti E, Malagoni AM, Gianesini S, Bartolomei I, Mascoli F, Salvi F. A prospective open-label study of endovascular treatment of chronic cerebrospinal venous insufficiency. J Vasc Surg. 2009 Dec;50(6):1348-58.e1-3. doi: 10.1016/j.jvs.2009.07.096. PMID 19958985
- [Derived] Zamboni P, Galeotti R, Salvi F, Giaquinta A, Setacci C, Alborino S, Guzzardi G, Sclafani SJ, Maietti E, Veroux P; Brave Dreams Research Group. Effects of Venous Angioplasty on Cerebral Lesions in Multiple Sclerosis: Expanded Analysis of the Brave Dreams Double-Blind, Sham-Controlled Randomized Trial. J Endovasc Ther. 2020 Feb;27(1):1526602819890110. doi: 10.1177/1526602819890110. Epub 2019 Nov 17. PMID 31735108
- [Derived] Zamboni P, Tesio L, Galimberti S, Massacesi L, Salvi F, D'Alessandro R, Cenni P, Galeotti R, Papini D, D'Amico R, Simi S, Valsecchi MG, Filippini G; Brave Dreams Research Group. Efficacy and Safety of Extracranial Vein Angioplasty in Multiple Sclerosis: A Randomized Clinical Trial. JAMA Neurol. 2018 Jan 1;75(1):35-43. doi: 10.1001/jamaneurol.2017.3825. PMID 29150995
- [Derived] Zamboni P, Bertolotto A, Boldrini P, Cenni P, D'Alessandro R, D'Amico R, Del Sette M, Galeotti R, Galimberti S, Liberati A, Massacesi L, Papini D, Salvi F, Simi S, Stella A, Tesio L, Valsecchi MG, Filippini G; Chair of the Steering Committee. Efficacy and safety of venous angioplasty of the extracranial veins for multiple sclerosis. Brave dreams study (brain venous drainage exploited against multiple sclerosis): study protocol for a randomized controlled trial. Trials. 2012 Oct 3;13:183. doi: 10.1186/1745-6215-13-183. PMID 23034121
- See also: Related Info — http://www.ospfe.it